CLINICAL TRIAL: NCT06117267
Title: A Single-arm, Single-center Clinical Study to Verify the Navigation Image Accuracy in Cervical Spine Surgery Using Anatase Spine Surgery Navigation System
Brief Title: Navigation Image Accuracy Test in Cervical Spine Surgery Using Anatase Spine Surgery Navigation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Di Chiu, Director, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMUH112-REC1-144
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cervical Spine Fusion
Keywords: Spine Surgery Navigation System
MeSH Terms: conditions — Klippel-Feil Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Anatase Spine Surgery Navigation System (Experimental): Using the navigation system during surgery
  Interventions: Device: Anatase Spine Surgery Navigation System

INTERVENTIONS:
Device: Anatase Spine Surgery Navigation System — Collect images with the probe touching the target position before screw implantation

SUMMARY:
The "Anatase" Spine Surgery Navigation System used in this study has obtained market approval in Taiwan(MOHW-MD-No.006663) and the United States (510(k) Numbers: K180523 and K220348).

The "Anatase" Spine Surgery Navigation System, also known as an Image Guide System, is indicated for precise positioning of surgical instruments or spinal implants, such as pedicle screw placement, during general spinal surgery. The system uses wireless optical tracking technology to track the position of instruments in relation to the surgical anatomy and register to the relative position in preoperative 3D CT imagery.

The aim of the study is to verify the accuracy of "Anatase" Spine Surgery Navigation System in Image-guided Cervical Spine Surgery. This trial will involve 8 subjects using the approved "Anatase" Spine Surgery Navigation System to collect images before screw implantation, and verify the accuracy of navigation images in cervical spine surgery.

DETAILED DESCRIPTION:
The "Anatase" Spine Surgery Navigation System, is composed of an Optical Tracker, Computer, No-Touch Reader and Dynamic Reference Frame (DRF). The Optical Tracker is a position sensor, it tracks the position of instruments with DRF by infrared light, allowing the instrument and vertebra to be positioned. The Computer is a touch screen panel PC running the proprietary spine NAVI software that guides the surgical procedure and display the results of the operation and computation. A No-Touch Reader, which attached on the Optical Tracker, is a no-touch sensor to identify instruments. It's a unique design and identification technology allows the instrument to be wirelessly identified, reducing the risk and time required to set up the instrument type. The system can track the position of patient's vertebra and instruments by mounting the DRF on patient's vertebra and instruments.

The "Anatase" Spine Surgery Navigation System is indicated for precise positioning of surgical instruments or spinal implants during general spinal surgery. The system helps to guide surgeons with real-time image and provides preoperative planning and intraoperative control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years
* Patients who need to undergo posterior cervical pedicle screw placement surgery
* The subject is willing to provide preoperative CT images and to use the navigation system during surgery for the verification of navigation image accuracy.
* Subjects are willing and able to comply with the procedures and requirements of this clinical trial.
* Subjects are able to understand and willing to sign the informed consent form.

Exclusion Criteria:

* Creutzfeldt-Jakob disease
* Known allergy to stainless steel
* Immunocompromised such as but not limited to Acquired Immunodeficiency Syndrome (AIDS), HIV infection, Severe Combined Immunodeficiency Syndrome, Thymic Hypoplasia
* Pregnant women
* Have a systematic or local infection, which may increase study risk
* Hereditary or acquired hemorrhagic diathesis or coagulation factor deficiency
* Use of anticoagulants
* Osteoporosis
* Be on uncontrolled diabetes mellitus.
* Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months.
* Previous history of cervical spine surgery
* Other medical conditions, as judged by a physician, may affect the physiological status for surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference between the actual and virtual (navigation system) distance of the probe. | during the surgery
  The assessor will measure the distance (mm) of the probe between the actual and virtual (navigation system) images.
Difference between the actual and virtual (navigation system) angle of the probe. | during the surgery
  The assessor will measure the angle (°) of the probe between the actual and virtual (navigation system) images.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Di Chiu, Principal Investigator — China Medical University Hospital